CLINICAL TRIAL: NCT02266394
Title: Hypoxia and Inflammatory Injury in Human Renovascular Hypertension : Phase 1 Trial of Mesenchymal Stem Cell Therapy
Brief Title: Hypoxia and Inflammatory Injury in Human Renovascular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Mississippi Medical Center (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stephen C. Textor, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-002799
Record Dates: First submitted 2014-09-18; First posted 2014-10-17 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Renal Artery Stenosis; Ischemic Nephropathy; Renovascular Disease; Chronic Kidney Disease
MeSH Terms: conditions — Renal Artery Obstruction; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell delivery (Active Comparator): To determine hemodynamic and immunologic changes associated with intra-renal delivery of adipose-derived MSC into human subjects with advanced RVD.
  Interventions: Drug: Mesenchymal stem cell
- Mesenchymal stem cell delivery with stent placement (Active Comparator): To test adjunctive delivery of MSC to individuals with advanced RVD undergoing renal artery stenting.
  Interventions: Drug: Mesenchymal stem cell; Procedure: Mesenchymal stem cell delivery with stent placement

INTERVENTIONS:
Drug: Mesenchymal stem cell — Intra-arterial infusion of the single-dose MSC
  Other Names: Mesenchymal stem cell delivery
Procedure: Mesenchymal stem cell delivery with stent placement — Intra-arterial stent placement after Mesenchymal stem cell infusion
  Arms: Mesenchymal stem cell delivery with stent placement

SUMMARY:
Current treatments for ARAS based on restoring blood flow alone have been unsuccessful at recovering kidney function. For this reason we are studying a stem cell product called "mesenchymal stem cells" or MSC. Mesenchymal stem cells (MSC) are grown from a person's own fat tissue (obtained as a fat biopsy) and infused back into the patient's own kidney.

This study is also being done to determine if the MSC infusion prior to percutaneous transluminal renal angioplasty with stenting (PTRA) further enhances changes in single kidney blood flow and restoration of kidney function, as well as to assess the relationship between MSC dose and measures of kidney function.

DETAILED DESCRIPTION:
These studies include participation by human subjects using a 3-day inpatient CRU protocol at St. Mary's Hospital. Studies include formal measurement of blood and urinary markers of kidney function, BOLD MR and multidetector CT scanning. Forty-two non-diabetic patients between 40 and 80 years of any race or ethnicity will be recruited. All will have hypertension (defined as BP≥140/90 mmHg or ongoing antihypertensive drug therapy) but will have less than 180 mmHg to be included (with or without drug therapy). These subjects will be free of cardiovascular events within 3 months and will not have implanted electrical devices, such as a pacemaker or defibrillator. All patients will have identified large vessel renovascular disease (RVD) for Aims 1, 2 and 3. At least 10% of these subjects will be of African-American descent (self-identified) and recruited in collaboration with the University of Mississippi under the direction of Dr. Luis Juncos and the University of Alabama under the direction of Dr. David Calhoun. For completion of Aims 2 and 3, a three-day evaluation will be repeated between three and four months later, and ongoing safety and imaging studies will be performed up to 24 months after MSC administration. Participants in these protocols will undergo transvenous kidney biopsy under the direction of Drs. McKusick and Misra and their colleagues in Interventional Radiology. All subjects for these studies will complete the research plan at Mayo Clinic, Rochester, Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine <2.2 mg/dL for Caucasian males, <2.0 Caucasian females,< 2.4 African-American males, <2.1 mg/dL African-American females
* Hypertension (Systolic BP>155 mm Hg) and/or requirement for two or more antihypertensive medications: no restrictions on antihypertensive agents, although loop diuretics will be changed to diluting site agents (e.g. hydrochlorothiazide, indapamide, metolazone) prior to study.
* Angiotensin Converting Enzyme (ACE inhibitor) or Angiotensin Receptor Blocker (ARB) therapy maintained or initiated at usual recommended daily dose (equivalent: 40 mg lisinopril) .

Exclusion Criteria:

* Diabetes requiring insulin or oral hypoglycemic medications (see text)
* Known allergy to furosemide or iodinated intravenous contrast
* Pregnancy
* Recent Cardiovascular event: Myocardial infarction, stroke, congestive heart failure within 3 months
* Cardiac ejection fraction less than 30%
* Evidence of hepatitis B or C, or HIV infection
* requirement for potentially nephrotoxic drugs, e.g. non-steroidal anti-inflammatory drugs
* Uncontrolled hypertension: SBP >180 mm Hg, despite antihypertensive therapy
* Kidney transplant
* Pacemaker, implantable defibrillator or other contraindication to Magnetic resonance imaging
* Inability to comply with breath-hold for 30 seconds
* History of deep venous thrombosis within 3 months of enrollment
* contraindications to renal biopsy including artificial valve requiring continuous anticoagulation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Kidney function | 3 months
  Renal Tissue oxygenation
Safety of Mesenchymal stem cell infusion | 2 years
  Number of patients with tissue injury markers

SECONDARY OUTCOMES:
Decrease in Kidney inflammation | 3 months
  Venous and tissue biomarkers of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Textor, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lerman LO. Cell-based regenerative medicine for renovascular disease. Trends Mol Med. 2021 Sep;27(9):882-894. doi: 10.1016/j.molmed.2021.06.004. Epub 2021 Jun 25. PMID 34183258
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials